CLINICAL TRIAL: NCT01533246
Title: A Phase 2 Study of OSI-906 in Patients With Asymptomatic or Mildly Symptomatic (Non-Opioid Requiring) Metastatic Castrate Resistant Prostate Cancer (CRPC)
Brief Title: Linsitinib in Treating Patients With Asymptomatic or Mildly Symptomatic Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00247; NCI-2012-00247 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000724845; CASE 6810 (Other: Case Comprehensive Cancer Center); 8872 (Other: CTEP); U01CA062502 (NIH)
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2013-12

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

ARMS (1):
- Treatment (linsitinib) (Experimental): Patients receive linsitinib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo serum and plasma sample collection at baseline, on day 1 of courses 2 and 4, and after completion of study treatment for correlative studies.
  Interventions: Drug: linsitinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: linsitinib — Oral Linsitinib 150mg, twice a day, days 1- 28
  Other Names: OSI-906
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well linsitinib works in treating patients with asymptomatic or mild symptomatic metastatic prostate cancer. Linsitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate time to prostate-specific antigen (PSA) progression based on Prostate Cancer Working Group (PCWG2) criteria.

II. To evaluate PSA response (proportion of patients achieving a PSA decline > 50% according to PCWG2 criteria in patients receiving linsitinib [OSI-906]).

III. To evaluate overall response rate (ORR) in patients with Response Evaluation Criteria in Solid Tumors (RECIST)-defined measurable disease receiving OSI-906.

SECONDARY OBJECTIVES:

I. To evaluate the effect of OSI-906 on time-to opiate use for cancer pain. II. To evaluate the effect of OSI-906 on radiographic progression-free survival (rPFS) of patients with asymptomatic or mildly symptomatic (non-opioid requiring) castrate-resistant prostate cancer (CRPC).

III. To evaluate the overall survival (OS) of patients with asymptomatic or mildly symptomatic (non-opioid requiring) CRPC receiving OSI-906.

IV. To further evaluate the safety of OSI-906 in patients with asymptomatic or mildly symptomatic (non-opioid requiring) CRPC.

TERTIARY OBJECTIVES:

I. To describe the effects of OSI-906 in the levels of androstenedione, dehydroepiandrostenedione (DHEA), DHEA-sulfate, p insulin-like growth factor-1 receptor (IGF-IR), and p-insulin receptor (IR). (Exploratory) II. To describe the effects of OSI-906 in the levels of transforming growth factor (TGF)-beta (b1), interleukin-6 (IL-6), tumor necrosis factor (TNF)-alpha (a), and monocyte chemotactic protein 1 (MCP-1) as markers of metastatic progression. (Exploratory) III. To describe the effects of OSI-906 on the number of circulating tumor cells (CTCs) and endothelial cells (CECs). (Exploratory) IV. To use ribonucleic acid (RNA) extracted from CTCs to evaluate effects on downstream targets of IGF-1R signaling after OSI-906 treatment. (Exploratory) V. To measure the effect of OSI-906 on the expression of IGF-1R on CTCs. (Exploratory)

OUTLINE:

Patients receive linsitinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo serum and plasma sample collection at baseline, on day 1 of courses 2 and 4, and after completion of study treatment for correlative studies.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM); if the patient is being treated with luteinizing hormone-releasing hormone (LHRH) agonists (patient who has not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to course 1 Day 1 and must be continued throughout the study
* Metastatic disease documented by positive bone scan or metastatic lesions other than liver or visceral metastasis on computed tomography (CT) or magnetic resonance imaging (MRI); if lymph node metastasis is the only evidence of metastasis, it must be ≥ 2 cm in diameter
* Prostate cancer progression documented by PSA according to PCWG2 or radiographic progression according to modified RECIST criteria
* Asymptomatic or mildly symptomatic from prostate cancer; a score of 0-1 on Brief Pain Inventory (BPI)-Short Form (SF) Question #3 (worst pain in last 24 hours) will be considered asymptomatic, and a score of 2-3 will be considered mildly symptomatic
* Patients who received combined androgen blockade or received second-line anti-androgen in the context of CRPC must have shown PSA progression after discontinuing the anti-androgen prior to enrollment (≥ 4 weeks since last flutamide, ≥ 6 weeks since last bicalutamide or nilutamide) and have progressive disease
* No patients with known brain metastases
* Understand and voluntarily sign an informed consent form
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Hemoglobin ≥ 10.0 g/dL independent of transfusion
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/μL
* Serum albumin ≥ 3.5 g/dL
* Serum creatinine < 1.5 times upper limit of normal (ULN) OR a calculated creatinine clearance ≥ 60 mL/min
* Serum potassium ≥ 3.5 mmol/L
* Serum bilirubin < 1.5 times ULN (except for patients with documented Gilbert's disease)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 times ULN
* Able to swallow the study drug
* Life expectancy of at least 6 months
* Men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* No history of clinically significant heart disease as evidenced by myocardial infarction or arterial thrombotic events in the past 6 months, severe or unstable angina, New York Heart Association (NYHA) Class II-IV heart disease, or cardiac ejection fraction measurement of < 50% at baseline
* No prolonged QTc > 470 msec (mean QTc with Bazett's correction) or history of familial long QT syndrome
* No other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 24 months
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-906
* No uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements
* Patients with insulin-dependent diabetes are excluded
* Patients with known history of HIV on combination antiretroviral therapy are ineligible
* Patients with known infectious hepatitis A, B, or C are ineligible
* No condition that, in the opinion of the investigator, would preclude participation in this trial
* See Disease Characteristics
* Prior therapy with ketoconazole and steroids is allowed provided patients have been off treatment for 4 weeks
* Prior investigational agents with novel adrenal inhibitors (i.e., Abiraterone or TAK700) are allowed provided these agents have been discontinued at least 4 weeks prior to enrollment
* Prior investigational agents with novel antiandrogens (i.e., MDV 3100) are allowed provided these agents have been discontinued at least 6 weeks prior to enrollment
* Prior therapy with Sipuleucel-T is allowed provided patients have documented evidence of disease progression as stated above
* Patients receiving any other hormonal therapy, including any dose of Megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), or any systemic corticosteroid must discontinue the agent for at least 4 weeks prior to enrollment; progressive disease (as defined above) must be documented after discontinuation of the hormonal therapy
* Patients on stable doses of bisphosphonates that show subsequent tumor progression may continue on this medication at the discretion of the treating physician; however, patients are not allowed to initiate bisphosphonate therapy within 4 weeks prior to starting therapy or throughout the study
* No prior systemic chemotherapy for CRPC; prior neoadjuvant and adjuvant chemotherapy are allowed when completed at least 12 months prior to enrollment
* No use of opiate analgesics for cancer-related pain, including codeine and dextropropoxyphene, currently or anytime within 4 weeks of Cycle 1 Day 1
* No prior use of IGF-1R inhibitors (monoclonal antibody or small molecule)
* No palliative radiation therapy to bone metastasis or radionuclide therapy for treatment of metastatic CRPC within 4 weeks of Cycle 1 Day 1
* Use of the potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine are prohibited

  * Other less potent CYP1A2 inhibitors/inducers are not excluded
* Supplements or complementary medicine/botanicals are not permitted while on protocol therapy, except for any combination of the following:

  * Conventional multivitamin supplements
  * Selenium
  * Lycopene
  * Soy supplements
* The use of concomitant steroids is not allowed unless patients are receiving physiological replacement disease for documented adrenal insufficiency
* Use of drugs that have a known risk of causing Torsades de Pointes (TdP) are prohibited within 14 days prior to study enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Barata P, Cooney M, Tyler A, Wright J, Dreicer R, Garcia JA. A phase 2 study of OSI-906 (linsitinib, an insulin-like growth factor receptor-1 inhibitor) in patients with asymptomatic or mildly symptomatic (non-opioid requiring) metastatic castrate resistant prostate cancer (CRPC). Invest New Drugs. 2018 Jun;36(3):451-457. doi: 10.1007/s10637-018-0574-0. Epub 2018 Feb 23. PMID 29476383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 patients were entered into the trial between February 2012 and April 2012 form local medical hospitals. One patient was considered ineligible and has been excluded from all analyses.
Groups:
- Treatment (Linsitinib): Patients receive linsitinib 150mg PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo serum and plasma sample collection at baseline, on day 1 of courses 2 and 4, and after completion of study treatment for correlative studies.
  linsitinib: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Linsitinib)
Started | 17
Completed | 15
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patients that received treatment.
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
Age, Customized [Number; unit: participants]
  50-59 years | 2
  60-69 years | 7
  70-79 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Analyzed Using the PCWG2 Definition
Description: Number of patients with a PSA Response will be evaluated according to the recommendations from National Cancer Institute Prostate-Cancer Working Group 2 (PCWG2) criteria. PSA decline of at least 50% from baseline confirmed by a second measurement at least 4 weeks later.
Time Frame: 12 weeks
Population: Patients that received treatment
Measure: Number; unit: participants
Groups:
- Treatment (Linsitinib): Patients receive linsitinib 150mg, PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo serum and plasma sample collection at baseline, on day 1 of courses 2 and 4, and after completion of study treatment for correlative studies.
  linsitinib: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
participants
  PSA Partial Response | 1
  PSA No Response | 16

2. Secondary Outcome: Incidence of Toxicities Based on CTCAE Version 4.0 Criteria
Description: Number of patients with at least possibly related to treatment toxicities grade 3 or higher based on Common Terminology Criteria for Adverse Events.
Time Frame: Up to 2 years
Population: Patients that received treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
participants | 1

3. Secondary Outcome: Number of Patients With Bidimensional Measurable Disease RECIST-based Response
Description: RECIST response categories: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: Up to 2 years
Population: Patients with soft tissue disease only
Measure: Number; unit: participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 10
participants
  Partial Response | 1
  Stable Disease | 8
  Progression | 1

4. Secondary Outcome: Time to PSA Progression (TTPP) Analyzed Using the PCWG2 Definition
Description: TTPP will be measured from protocol registration to appearance of PSA progression as defined by the criteria of the PSA Working Group response criteria. The end point for progression will be calculated at the time a 25% increase in PSA has been achieved.
Time Frame: assessed up to 12 weeks
Population: Patients that received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
months | 1.8 [0.9 to 2.8]

5. Secondary Outcome: Overall Survival Based on the RECIST v1.1
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Up to 2 years
Population: Patients that received treatment
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
Months | 3.7 [3 to 6.7]

6. Secondary Outcome: Progression Free Survival
Description: Progression Free survival (PFS) time was measured as the time from the date of on study up to the date of occurrence of the first event defining a disease progression or death due to any cause, whichever occurred first.
Time Frame: assessed up to 2 years
Population: Patients that received treatment
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
Months | 4.7 [3 to 6.7]

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events from start of treatment to 30 days after treatment up to a period of 6 months
Arm/Group | Treatment (Linsitinib)
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Linsitinib) (N=17)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Linsitinib) (N=17)
Aspartate aminotransferase increased (Investigations) | 11 (15)
Creatinine increased (Investigations) | 8 (12)
Alanine aminotransferase increased (Investigations) | 7 (8)
Lymphocyte count decreased (Investigations) | 6 (10)
Electrocardiogram QT corrected interval prolonged (Investigations) | 5 (8)
Platelet count decreased (Investigations) | 3 (3)
Weight loss (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (5)
Neutrophil count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (18)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 10 (16)
Non-cardiac chest pain (General disorders) | 3 (3)
Irritability (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral thigh cramps intermittent (Musculoskeletal and connective tissue disorders) | 1 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 4 (5)
Upper respiratory infection (Infections and infestations) | 2 (2)
Renal calculi (Renal and urinary disorders) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (2)
Penile hemorrhage (Reproductive system and breast disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less